CLINICAL TRIAL: NCT04817072
Title: Evaluation of Mood Disorders Under Biologics (Anti-TNF Alpha) in Chronic Inflammatory Rheumatic Disease
Brief Title: Evaluation of Mood Disorders Under Biologics in Chronic Inflammatory Rheumatic Disease
Acronym: EMOTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P/2019/462
Record Dates: First submitted 2021-01-29; First posted 2021-03-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-11

CONDITIONS: Rheumatic Diseases; Mood Disorders
Keywords: TNF alpha inhibitor
MeSH Terms: conditions — Rheumatic Diseases; Mood Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic inflammatory rheumatic disease (Other): Patients presenting a chronic inflammatory rheumatic disease (rheumatoid arthritis, spondyloarthritis or psoriatic arthritis), requiring anti-TNFa therapy and with a QIDS SR-16 (QIDS-SR 16-Quick Inventory of Depressive Symptomatology-Self Reported 16 items) score between 6 and 19
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample (20mL) for pro-inflammatory cytokines assay

SUMMARY:
Chronic inflammatory rheumatic diseases (CIRD) affect many organ systems. Painful sensations within the joints spine, hand and foot deformities, low quality of life and psychosocial status in patients with rheumatoid arthritis, spondyloarthritis and psoriatic arthritis can lead to the development of anxiety and depression. Prevalences of anxiety increase in patients suffering of CIRD, compared with healthy individuals. Another connection has been identified by the links between depression and systemic inflammation. It is proven that higher plasma levels of pro-inflammatory cytokines such as tumor necrosis factor alpha (TNFa) affect neurotransmitter metabolism, with influence on patients mood. The purpose of EMOTION study is therefore to analyze thymic variation under TNFa therapy, as treatment of CIRDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 ; ≤ 80)
* Patient with rheumatoid arthritis (RA) according to the ACR 2010 criteria, axial or peripheral spondyloarthritis (SpA) according to ASAS criteria, ankylosing spondylitis (AS) according to the New York criteria or psoriatic arthritis (PsA) according to CASPAR criteria
* Signature of informed consent
* Affiliation to a French social security or receiving such a scheme

Exclusion Criteria:

* Patient having previously received anti-TNFα treatment
* Patient with previously diagnosed depressive or psychiatric pathology and / or receiving anti-depressant treatment
* Subjects with limited legal capacity.
* Subjects judged by the investigator to be unlikely to comply with study procedures
* Subjects with no social security coverage.
* Pregnant women.
* Subjects still in the exclusion period of another study, or according to the national registry of clinical trial participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Severity of depressive symptoms | 1 month after initiation of anti-TNFa therapy
  Score achieved on the validated self-report questionnaire (QIDS SR16) evaluating the severity of depressive symptoms

SECONDARY OUTCOMES:
Evaluation of disease activity | 3 months after initiation of anti-TNFa therapy
  Evaluation with CPDAI (Composite Psoriatic Disease Activity Index) (minimum value: 0; maximum value: 15; increases with the activity of the disease)
Evaluation of disease activity | 3 months after initiation of anti-TNFa therapy
  Evaluation with DAS28 (Disease Activity Score 28-joint count) (minimum value: 0; maximum value: 9.4; increases with the activity of the disease)
Evaluation of disease activity | 3 months after initiation of anti-TNFa therapy
  Evaluation with BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) (minimum value: 0 (no disease activity); maximum value: 10 (very active disease))
Evaluation of disease activity | 3 months after initiation of anti-TNFa therapy
  Evaluation with ASDAS (Ankylosing Spondylitis Disease Activity Score) (minimum value: 0 (no disease activity); value >3.5 between : very high disease activity)
Evaluation of Fatigue | 3 months after initiation of anti-TNFa therapy
  Evaluation with Functional Assessment of Chronic Illness Therapy
Evaluation of Pleasure | 3 months after initiation of anti-TNFa therapy
  Evaluation with Snaith-Hamilton pleasure scale (minimum value: 0 (no disease activity); maximum value: 14 (very active disease)). A higher total SHAPS score indicated higher levels of anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Toussirot, PU-PH, Principal Investigator — Besançon University Hospital
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No